CLINICAL TRIAL: NCT00333138
Title: Double-blind, Randomized, Placebo-controlled, Parallel-group, Multicenter Study Evaluating the Safety, Tolerability and Effect on MRI Lesion Parameters of FTY720 vs Placebo in Patients With Relapsing Multiple Sclerosis Including 18 Month Extension Phase
Brief Title: Efficacy and Safety of FTY720 in Patients With Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720D2201; CFTY720D2201E1 (Other: Novartis); NCT00235430 (obsolete NCT alias)
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
Keywords: FTY720; MS; Multiple Sclerosis; RRMS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Fingolimod (FTY720) 1.25 mg/day (Experimental): Core study: patients received fingolimod 1.25 mg, once daily for 6 months. Extension: In dose -blind period and open label, fingolimod 1.25 mg once daily for 9-18 months (6 months to 24 months). Later, all patients converted to fingolimod 0.5 mg, once daily for rest of the study participation.
  Interventions: Drug: FTY720
- Placebo/Fingolimod (FTY720) (Placebo Comparator): Core study: patients received placebo, once daily for 6 months. Extension: In dose-blind period patients were re-randomized into either fingolimod 1.25 mg or 5.0 mg once per day for 6-15 months. In open-label period patients received fingolimod 1.25 mg once per day for 15 to 24 months. Later, all patients converted to fingolimod 0.5 mg, once daily for rest of the study participation.
  Interventions: Drug: Placebo
- Fingolimod (FTY720) 5.0 mg/day (Experimental): Core study: patients received fingolimod 5.0 mg, once daily for 6 months. Extension: In dose-blind period fingolimod 5.0 mg once daily for 6-15 months. For open-label phase 15 to 24 months 1.25mg once daily. Later, all patients converted to fingolimod 0.5 mg, once daily for rest of the study participation.
  Interventions: Drug: FTY720

INTERVENTIONS:
Drug: FTY720 — FTY720 capsule was taken orally once a day
  Arms: Fingolimod (FTY720) 1.25 mg/day; Fingolimod (FTY720) 5.0 mg/day
Drug: Placebo — Placebo 1.25 mg capsule was given once daily
  Arms: Placebo/Fingolimod (FTY720)

SUMMARY:
This study evaluated the safety, tolerability and effect on MRI lesion parameters of FTY720 in patients with relapsing multiple sclerosis.

ELIGIBILITY:
Core Study

Inclusion Criteria:

* Diagnosis of relapsing multiple Sclerosis (MS)
* Patients with at least two documented relapses in the previous 2 years or one documented relapse in the last year
* Patients with an Expanded Disability Status Scale (EDSS) score of 0-6

Extension Study

* A positive Gd-enhanced MRI scan at screening (in case the first MRI scan obtained at screening was negative, a second scan could have been obtained 1 month later)
* Neurologically stable with no evidence of relapse within 30 days prior to randomization,or during the Screening and Baseline periods.
* Female patients either post-menopausal, surgically incapable of bearing children, or practicing an acceptable method of birth control. Females of childbearing potential with a negative pregnancy test at baseline prior to entry into the treatment period.

Exclusion Criteria:

Core Study

* Patients with other chronic disease of the immune system, malignancies, pulmonary or heart disease, etc
* Pregnant or nursing women

Extension Study

* Patients who had permanently discontinued study drug prior to the Month 6 visit of the core study
* Patients with diabetes mellitus (to reduce the risk of ME), and therefore ongoing patients with diabetes mellitus or who developed diabetes mellitus were discontinued from the study)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 281 (Actual)
Dates: Start 2003-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (26):
- Canada (4):
  - Novartis Investigational site, Montreal
  - Novartis Investigational site, Ottawa
  - Novartis Investigational site, Toronto
  - Novartis Investigational site, Vancouver
- Novartis Investigational site, Copenhagen, Denmark
- Finland (2):
  - Novartis Investigational site, Helsinki
  - Novartis Investigational site, Turku
- France (2):
  - Novartis Investigational site, Lille
  - Novartis Investigational site, Marseille
- Germany (2):
  - Novartis Investigational site, Schwendi
  - Novartis Investigational site, Würzburg
- Italy (4):
  - Novartis Investigational site, Gallarate
  - Novartis Investigational site, Genova
  - Novartis Investigational site, Milan
  - Novartis Investigational site, Roma
- Novartis Investigational site, Warsaw, Poland
- Portugal (2):
  - Novartis Investigational site, Coimbra
  - Novartis Investigational site, Lisbon
- Spain (5):
  - Novartis Investigational site, Barcelona
  - Novartis Investigational site, Madrid
  - Novartis Investigational site, Málaga
  - Novartis Investigational site, Seville
  - Novartis Investigational site, Valencia
- Switzerland (2):
  - Novartis Investigational site, Basel
  - Novartis Investigational site, Zurich
- Novartis Investigational site, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Zarbin MA, Jampol LM, Jager RD, Reder AT, Francis G, Collins W, Tang D, Zhang X. Ophthalmic evaluations in clinical studies of fingolimod (FTY720) in multiple sclerosis. Ophthalmology. 2013 Jul;120(7):1432-9. doi: 10.1016/j.ophtha.2012.12.040. Epub 2013 Mar 24. PMID 23531349
- [Derived] Kappos L, Antel J, Comi G, Montalban X, O'Connor P, Polman CH, Haas T, Korn AA, Karlsson G, Radue EW; FTY720 D2201 Study Group. Oral fingolimod (FTY720) for relapsing multiple sclerosis. N Engl J Med. 2006 Sep 14;355(11):1124-40. doi: 10.1056/NEJMoa052643. PMID 16971719

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Core study: patients received placebo, once daily for 6 months. Extension: In dose-blind period patients were re-randomized into either fingolimod 1.25 mg or 5.0 mg once per day for 6-15 months. In open-label period patients received fingolimod 1.25 mg once per day for 15 to 24 months. Later, all patients converted to fingolimod 0.5 mg, once daily for rest of the study participation.
- Fingolimod (FTY720) 5.0 mg/Day: Core study: patients received fingolimod 5.0 mg, once daily for 6 months. Extension: In dose-blind period fingolimod 5.0 mg once daily for 6-15 months. For open-label phase 1.25mg once daily for 15 to 24 months. Later, all patients converted to fingolimod 0.5 mg, once daily for rest of the study participation.
Period: Core Study (6 Months)
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Started | 93 | 94 | 94
Completed | 86 | 88 | 82
Not Completed | 7 | 6 | 12
Not completed — Adverse Event | 4 | 5 | 8
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Laboratory abnormality | 0 | 0 | 1
Period: Extension Study (Month6 to End of Study)
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Started | 83 | 87 | 80
Completed | 40 | 45 | 37
Not Completed | 43 | 42 | 43
Not completed — Abnormal laboratory value | 3 | 2 | 2
Not completed — Administrative problems | 1 | 1 | 2
Not completed — Adverse Event | 15 | 19 | 15
Not completed — Protocol Violation | 0 | 0 | 3
Not completed — Withdrawal by Subject | 14 | 13 | 14
Not completed — Lack of Efficacy | 7 | 4 | 7
Not completed — Patient no longer required study drug | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day | Total
Number analyzed (Participants) | 93 | 94 | 94 | 281
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (8.80) | 38.1 (9.54) | 38.3 (10.51) | 37.8 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 71 | 66 | 199
  Male | 31 | 23 | 28 | 82

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Gadolinium (Gd)-Enhanced T1-weighted Lesions at Month 6 (Core)
Description: Total number of post-baseline Gd-enhanced lesions is calculated as a sum of all Gd-enhanced lesions seen on post-baseline scans per visit. Real (not per slice) lesions are counted in this analysis.
Time Frame: Month 6 (Core)
Population: All randomized patients who received at least 1 dose of study drug during the core study were included in the ITT population. Number of patients with T1 information recorded at scan were included in the analysis.
Measure: Mean (Standard Deviation); unit: GD- enhanced T1 lesions
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 83 | 90 | 87
GD- enhanced T1 lesions | 2.3 (4.23) | 1.4 (5.69) | 0.4 (0.82)

2. Secondary Outcome: Percentage of Participants Free of T1-weighted Lesions
Description: A patient was defined as free of lesions if s/he had zero lesions. The last observation was the last observation available for each patient which ranged from 1 to 2801 days
Time Frame: Baseline, Months 6 (core), 12, 60 and Last Observation (up to 80 months in average)
Population: All randomized patients who received at least 1 dose of study drug during the core study were included in the ITT population. Number of patients with T1 information recorded at scan were included in the analysis. The "n" in each category indicates number of patients wih information recorded at scan
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 93 | 94 | 94
percentage of participants
  Baseline (Core) n=93, 92, 93 | 49.5 | 52.2 | 48.4
  Month 6 (Core) n= 83, 90, 87 | 47.0 | 76.7 | 78.2
  Month 12 (Extension) n= 72, 77, 71 | 79.2 | 83.1 | 88.7
  Month 60 (Extension) n= 45, 49, 44 | 91.1 | 91.8 | 93.2
  Last observation (Extension) n= 92, 93, 92 | 81.5 | 83.9 | 83.7

3. Primary Outcome: Mean Number of Gadolinium (Gd)-Enhanced T1-weighted Lesions at Month 12
Description: as for outcome 1
Time Frame: Month 12 (extension)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: GD- enhanced T1 lesions
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 72 | 77 | 71
GD- enhanced T1 lesions | 0.4 (0.95) | 1.0 (5.81) | 0.2 (0.47)

4. Primary Outcome: Mean Number of Gadolinium (Gd)-Enhanced T1-weighted Lesions at Month 60
Description: as for outcome 1
Time Frame: Month 60 (extension)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: GD- enhanced T1 lesions
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 45 | 49 | 44
GD- enhanced T1 lesions | 0.2 (0.7) | 0.2 (0.92) | 0.1 (0.55)

5. Primary Outcome: Mean Number of Gadolinium (Gd)-Enhanced T1-weighted Lesions at End of Study
Description: Total number of post-baseline Gd-enhanced lesions is calculated as a sum of all Gd-enhanced lesions seen on post-baseline scans per visit. Real (not per slice) lesions are counted in this analysis. The last observation was the last observation available for each patient which ranged from 1 to 2801 days
Time Frame: Last observation (Up to 80 months in average)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: GD- enhanced T1 lesions
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 92 | 93 | 92
GD- enhanced T1 lesions | 0.8 (2.87) | 0.4 (1.39) | 0.5 (1.65)

6. Secondary Outcome: Percentage of Patients Free of Gd-enhanced T1-weighted and New T2- Weighted Lesions by Visit
Description: A patient was defined as free of lesions if s/he had zero lesions. The sum of all new T2-weighted lesions at Month 1 to last observation was zero (the sum is missing if one of the assessments was missing). New T2 lesions at a specific visit were assessed relative to the previous visit scan. Exception: new T2 lesions at Month 24 were assessed relative to Month 12. The last observation was the last observation available for each patient which ranged from 1 to 2801 days
Time Frame: Month 6 and 12, 60, last observation (up to 80 months in average)
Population: All randomized patients who received at least 1 dose of study drug during core study were included in the ITT population. The "n" number of patients with T2 and T1 information recorded at scan
Measure: Number; unit: percentage of paticipants
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 93 | 94 | 94
percentage of paticipants
  Month 6 (Core), n= 80, 87, 83 | 47.5 | 77.0 | 80.7
  Month 12 (Extension) n=70, 77, 70 | 57.1 | 67.5 | 72.9
  Month 60 (Extension) n=45, 49, 43 | 88.9 | 87.8 | 83.7
  Last observation (Extension) n=92, 93,90 | 72.8 | 76.3 | 78.9

7. Secondary Outcome: Mean Number of New T2-weighted Lesions
Description: New T2 lesions at a specific visit were assessed relative to the previous visit scan. The total number of lesions (Month 1 to end of study) is calculated as the sum of the number of lesions at Months 1 to 6, Month 12, Month 60 and last observation. The last observation was the last observation available for each patient which ranged from 1 to 2801 days
Time Frame: (Core) Month 6 and (Extension) 12, 60, last observation (up to 80 months in average)
Population: All randomized patients who received at least 1 dose of study drug during the core study were included in the ITT population. The "n" in each category indicates participants with T2 information recorded at specific timepoints
Measure: Mean (Standard Deviation); unit: GD enhanced T2 lesions
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 93 | 94 | 94
GD enhanced T2 lesions
  Month 6 (Core), n= 82,88, 84 | 1.0 (2.37) | 0.5 (2.07) | 0.1 (0.34)
  Month 12 (Extension) n=71, 79, 71 | 0.8 (1.41) | 1.4 (5.56) | 0.6 (1.10)
  Month 60 (Extension) n=45, 50, 43 | 0.4 (1.25) | 0.5 (1.36) | 0.3 (0.97)
  Last observation (Extension) n=92, 93, 91 | 0.7 (1.99) | 0.6 (1.51) | 0.5 (1.64)

8. Secondary Outcome: Volume of T2-weighted Lesions
Description: Volume of total T2-weighted lesions by visit were summarized. The last observation was the last observation available for each patient which ranged from 1 to 2801 days
Time Frame: (Core) Month 6 and (Extension) 12, 60, last observation (up to 80 months in average)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 93 | 94 | 94
mm^3
  Month 6 (Core) n=85, 91, 87 | 9016.0 (10361.83) | 10084.6 (14774.16) | 8331.1 (10162.01)
  Month 12 (Extension) n= 73, 79, 72 | 8264.1 (10121.43) | 10707.1 (14887.66) | 8363.2 (10694.82)
  Month 60 (Extension) n=45, 50, 44 | 6698.3 (9569.98) | 9498.7 (9765.60) | 6626.9 (9146.01)
  Last observation (Extension) n=87, 91, 88 | 8757.2 (10127.01) | 10090.2 (13999.50) | 8061.8 (9003.47)

9. Secondary Outcome: Change From Baseline in Volume of Total T2-weighted Lesions
Description: Change in volume of total T2-weighted lesions by visit were summarized. Negative values indicate improvement (reduction in lesion volume) and positive values worsening (increase in lesion volume). The last observation was the last observation available for each patient which ranged from 1 to 2801 days.
Time Frame: Baseline to month 6, 12, 60 and Last observation (up to 80 months in average)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 93 | 94 | 94
mm^3
  Month 6 (core) n=85, 89, 86 | 146.15 (1683.602) | -115.81 (1031.799) | -607.97 (1705.486)
  Month 12 (extension) n=73, 77, 71 | 144.96 (1513.577) | 1.66 (1714.731) | -513.35 (1943.338)
  Month 60 (extension) n=45, 49, 43 | -621.82 (1338.966) | -204.09 (2238.182) | -1429.98 (3928.944)
  Last observation (extension) n= 87, 89, 87 | -178.86 (1884.904) | -92.24 (3033.041) | -907.48 (2997.668)

10. Secondary Outcome: Time to Event Analysis: Kaplan Meier Estimates of Percentage of Relapse-free Patients
Description: The Expanded Disability Status Scale (EDSS) is a scale for assessing disability in 8 functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, other functions). An overall score ranging from 0 (normal) to 10 (death due to MS) is calculated. Disability progression was determined by the EDSS score based on the following criteria: One point increase from baseline in patients with baseline EDSS score from 0 to 5.0; or half a point increase in patients with baseline EDSS score of 5.5 or above. Percent of patients free of disability progression was calculated using the Kaplan-Meier method. The last observation was the last observation available for each patient which ranged from 1 to 2801 days
Time Frame: Month 6,12,60 and Last observation (up to 80 months in average)
Population: All randomized patients who received at least 1 dose of study drug during the core study were included in the ITT population. A patient at risk are those continuing in the study without an event before the specified timepoint The "n" denotes number of patients at risk.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg/Day | Fingolimod (FTY720) 5.0 mg/Day
Number analyzed (Participants) | 93 | 94 | 94
percentage of participants
  0 days (n=93,94,94) | 1.00 [1.000 to 1.000] | 1.00 [1.000 to 1.000] | 1.00 [1.000 to 1.000]
  200 days (n=57, 73, 70) | 0.69 [0.589 to 0.782] | 0.86 [0.786 to 0.929] | 0.86 [0.782 to 0.928]
  400 days (n=48, 63, 60) | 0.62 [0.520 to 0.725] | 0.78 [0.699 to 0.871] | 0.79 [0.707 to 0.878]
  600 days (n=41, 57, 52) | 0.58 [0.478 to 0.688] | 0.76 [0.669 to 0.849] | 0.78 [0.690 to 0.867]
  800 days (n=38, 48, 48) | 0.55 [0.477 to 0.662] | 0.75 [0.652 to 0.838] | 0.75 [0.653 to 0.843]
  1000 days (n=35, 42, 45) | 0.53 [0.416 to 0.634] | 0.70 [0.595 to 0.798] | 0.75 [0.653 to 0.843]
  1200 days (n=30, 38 40) | 0.51 [0.399 to 0.619] | 0.66 [0.55 to 0.770] | 0.70 [0.594 to 0.802]
  1400 days (n=29, 36, 35) | 0.51 [0.399 to 0.619] | 0.63 [0.516 to 0.739] | 0.70 [0.594 to 0.802]
  1600 days (n=27, 34, 34) | 0.51 [0.399 to 0.619] | 0.61 [0.496 to 0.724] | 0.68 [0.570 to 0.786]
  1800 days (n=25, 33, 33) | 0.51 [0.399 to 0.619] | 0.61 [0.496 to 0.724] | 0.68 [0.570 to 0.786]
  2000 days (n=23, 31, 31) | 0.51 [0.399 to 0.619] | 0.59 [0.475 to 0.707] | 0.66 [0.545 to 0.769]
  2200 days (n=22, 28, 30) | 0.49 [0.373 to 0.600] | 0.55 [0.433 to 0.673] | 0.66 [0.545 to 0.769]
  2400 days (n=21, 26, 27) | 0.46 [0.348 to 0.581] | 0.55 [0.433 to 0.673] | 0.66 [0.545 to 0.769]
  2600 days (n=9, 12, 12) | 0.44 [0.313 to 0.558] | 0.55 [0.433 to 0.673] | 0.66 [0.545 to 0.769]
  2880 days (n=0, 0, 0) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

11. Secondary Outcome: Mean Trough Blood Concentrations of FTY720
Description: For each patient, the arithmetic mean of the two FTY720 trough blood levels from month 3 and 6 was calculated. This was taken as the patient's steady-state trough levels. Venous blood samples (3 mL) were collected before the dose in ethylenediaminetetraacetic acid (EDTA)-containing tubes at protocol-scheduled visits at months 3 and 6 in all patients.
Time Frame: Month 3 and 6
Population: Pharmacokinetics population included all the patients who had sample collected and analysis was performed
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- FTY720 1.25 mg/Day: Patients randomized to fingolimod 1.25 mg/d in the core study who received fingolimod 1.25 mg/d in the dose-blind period of the extension study and initially in the open-label period and were later converted to fingolimod 0.5 mg/d.
- FTY720 5.0 mg/Day: Patients randomized to fingolimod 5.0 mg/d in the core study who received fingolimod 5.0 mg/d in the dose-blind period of the extension study. All patients received fingolimod 1.25 mg/d initially in the open-label period and were later converted to fingolimod 0.5 mg/d.
Arm/Group | FTY720 1.25 mg/Day | FTY720 5.0 mg/Day
Number analyzed (Participants) | 68 | 56
ng/mL
  Month 3 (core) | 7.64 (5.44) | 30.5 (18.8)
  Month 6 (core) | 7.38 (4.57) | 28.9 (22.1)

ADVERSE EVENTS:
Groups:
- Fingolimod (FTY720) 1.25 mg: Core study: patients received fingolimod 1.25 mg, once daily for 6 months. Extension: In dose -blind period and open label, fingolimod 1.25 mg once daily for 9-18 months (6 months to 24 months). Later, all patients converted to fingolimod 0.5 mg, once daily for rest of the study participation.
- Fingolimod (FTY720) 5.0 mg: Core study: patients received fingolimod 5.0 mg, once daily for 6 months. Extension: In dose-blind period fingolimod 5.0 mg once daily for 6-15 months. For open-label phase 1.25mg once daily for 15 to 24 months. Later, all patients converted to fingolimod 0.5 mg, once daily for rest of the study participation.
Arm/Group | Placebo | Fingolimod (FTY720) 1.25 mg | Fingolimod (FTY720) 5.0 mg
Serious Adverse Events (participants affected / at risk) | 25/93 | 19/94 | 32/94
Other Adverse Events (participants affected / at risk) | 86/93 | 88/94 | 92/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=93) | Fingolimod (FTY720) 1.25 mg (N=94) | Fingolimod (FTY720) 5.0 mg (N=94)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 3
Coronary artery thrombosis (Cardiac disorders) | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Adrenal mass (Endocrine disorders) | 0 | 0 | 1
Eye oedema (Eye disorders) | 1 | 0 | 0
Macular oedema (Eye disorders) | 0 | 2 | 2
Retinal detachment (Eye disorders) | 1 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 2
Concomitant disease progression (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 1 | 0
Heart rate abnormal (Investigations) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 1 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Varicose ulceration (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=93) | Fingolimod (FTY720) 1.25 mg (N=94) | Fingolimod (FTY720) 5.0 mg (N=94)
Leukopenia (Blood and lymphatic system disorders) | 7 | 14 | 15
Lymphopenia (Blood and lymphatic system disorders) | 13 | 18 | 18
Palpitations (Cardiac disorders) | 5 | 1 | 3
Conjunctivitis (Eye disorders) | 2 | 7 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 6 | 10 | 8
Aphthous stomatitis (Gastrointestinal disorders) | 4 | 5 | 4
Constipation (Gastrointestinal disorders) | 12 | 4 | 12
Diarrhoea (Gastrointestinal disorders) | 12 | 18 | 15
Dyspepsia (Gastrointestinal disorders) | 4 | 10 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 1 | 1
Nausea (Gastrointestinal disorders) | 8 | 10 | 16
Toothache (Gastrointestinal disorders) | 2 | 5 | 8
Vomiting (Gastrointestinal disorders) | 5 | 6 | 6
Asthenia (General disorders) | 8 | 4 | 3
Chest pain (General disorders) | 2 | 4 | 5
Fatigue (General disorders) | 22 | 23 | 16
Gait disturbance (General disorders) | 2 | 5 | 2
Oedema peripheral (General disorders) | 5 | 5 | 5
Pyrexia (General disorders) | 6 | 6 | 12
Bronchitis (Infections and infestations) | 9 | 17 | 12
Cystitis (Infections and infestations) | 4 | 2 | 6
Ear infection (Infections and infestations) | 1 | 6 | 3
Gastroenteritis (Infections and infestations) | 4 | 8 | 14
Herpes zoster (Infections and infestations) | 4 | 7 | 4
Influenza (Infections and infestations) | 16 | 23 | 22
Nasopharyngitis (Infections and infestations) | 34 | 39 | 42
Oral herpes (Infections and infestations) | 5 | 5 | 4
Pharyngitis (Infections and infestations) | 7 | 11 | 5
Respiratory tract infection (Infections and infestations) | 2 | 5 | 3
Rhinitis (Infections and infestations) | 6 | 5 | 2
Sinusitis (Infections and infestations) | 10 | 12 | 12
Tooth abscess (Infections and infestations) | 1 | 6 | 3
Tooth infection (Infections and infestations) | 2 | 7 | 7
Upper respiratory tract infection (Infections and infestations) | 19 | 19 | 18
Urinary tract infection (Infections and infestations) | 11 | 10 | 11
Viral upper respiratory tract infection (Infections and infestations) | 5 | 6 | 4
Contusion (Injury, poisoning and procedural complications) | 6 | 5 | 4
Fall (Injury, poisoning and procedural complications) | 7 | 6 | 4
Joint sprain (Injury, poisoning and procedural complications) | 4 | 5 | 2
Alanine aminotransferase increased (Investigations) | 18 | 12 | 15
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 2
Lymphocyte count decreased (Investigations) | 3 | 6 | 7
White blood cell count decreased (Investigations) | 4 | 5 | 5
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 6 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 14 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 16 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 4 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 15 | 15
Tendonitis (Musculoskeletal and connective tissue disorders) | 7 | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5 | 5
Dizziness (Nervous system disorders) | 13 | 8 | 10
Headache (Nervous system disorders) | 28 | 35 | 25
Hypoaesthesia (Nervous system disorders) | 13 | 8 | 9
Migraine (Nervous system disorders) | 10 | 6 | 6
Muscle spasticity (Nervous system disorders) | 1 | 2 | 6
Paraesthesia (Nervous system disorders) | 9 | 10 | 5
Somnolence (Nervous system disorders) | 1 | 4 | 6
Tremor (Nervous system disorders) | 3 | 5 | 2
Anxiety (Psychiatric disorders) | 4 | 7 | 7
Depression (Psychiatric disorders) | 15 | 12 | 14
Insomnia (Psychiatric disorders) | 12 | 15 | 8
Pollakiuria (Renal and urinary disorders) | 5 | 3 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 9 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 5 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 16 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 9
Acne (Skin and subcutaneous tissue disorders) | 3 | 3 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7 | 6
Eczema (Skin and subcutaneous tissue disorders) | 3 | 6 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 7 | 6 | 8
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 0 | 1
Hypertension (Vascular disorders) | 13 | 19 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.